CLINICAL TRIAL: NCT05162768
Title: A Phase 3 Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Daily Subcutaneous Injections of Elamipretide in Subjects With Primary Mitochondrial Disease Resulting From Pathogenic Nuclear DNA Mutations (nPMD) NuPower
Brief Title: Study to Evaluate Efficacy and Safety of Elamipretide in Subjects With Primary Mitochondrial Disease From Nuclear DNA Mutations (nPMD)
Acronym: NuPower
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIMD-301
Record Dates: First submitted 2021-12-08; First posted 2021-12-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Mitochondrial Myopathies; Mitochondrial Pathology; Mitochondrial DNA Mutation; Mitochondrial Diseases; Mitochondrial DNA Deletion; Mitochondrial DNA Depletion; Mitochondrial Metabolism Defect; Mitochondrial Complex I Deficiency
Keywords: primary mitochondrial myopathy (PMM); nuclear DNA mutations n(PMD); exercise intolerance; muscle weakness; mitochondrial dysfunction; POLG; TWINKLE; progressive external ophthalmoplegia; Elamipretide; mitochondrial replisome; replisome related mutations; MTP-131; primary mitochondrial disease (PMD)
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases; Mitochondrial complex I deficiency; Muscle Weakness; Ophthalmoplegia, Chronic Progressive External | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Intervention Model Description: In this 48-week trial, subjects will be randomized (in a ratio of 1:1) to one of two groups: single daily subcutaneous doses of 60mg elamipretide, or, matching placebo, using a central randomization stratified by whether or not subjects have nPMD associated with replisome-related mutations.
  130 subjects, consisting of 90 subjects with nPMD associated mutations of the mitochondrial replisome for primary analysis and an additional subset of up to 40 subjects who have nPMD associated with other non-replisome-related pathogenic mutations specific to nuclear DNA. Three periods: Screening (up to 28 days), Treatment (48 Weeks) and Follow-Up Period (4 weeks).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial personnel and subjects will be blinded to treatment until the database is locked. The Investigator will contact the Sponsor prior to unblinding any subject's treatment sequence unless in the instance of a medical emergency.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elamipretide (Experimental): 0.75 mL of 80mg/mL solution of elamipretide for a single daily SC dose of 60mg elamipretide
  Interventions: Drug: Elamipretide
- Placebo (Placebo Comparator): 0.75 mL of 80mg/mL solution of matching placebo for a single daily SC dose of 60mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elamipretide — 60 mg of elamipretide administered as once daily 0.75 mL subcutaneous injections for 48 weeks
  Other Names: MTP-131
  Arms: Elamipretide
Drug: Placebo — Placebo administered as once daily 0.75 mL subcutaneous injections for 48 weeks
  Arms: Placebo

SUMMARY:
SPIMD-301 is a 48-week, randomized, double-blind, parallel-group, placebo-controlled trial to assess efficacy and safety of single daily subcutaneous (SC) administration of elamipretide as a treatment for subjects with primary mitochondrial myopathy associated with nuclear DNA mutations (nPMD).

DETAILED DESCRIPTION:
This 48-week randomized, double-blind, parallel-group, placebo-controlled trial will enroll approximately 130 subjects, consisting of 90 subjects who have nPMD associated with pathogenic mutations of the mitochondrial replisome("replisome-related mutations") for primary analysis and an additional subset of up to 40 subjects who have nPMD associated with other non-replisome-related pathogenic mutations specific to the nuclear DNA. Efficacy and safety of single daily SC doses of elamipretide administered as a treatment for subjects who have primary mitochondrial myopathy associated with nPMD will be determined. Subjects will be randomized 1:1 to 60mg Elamipretide or matching placebo groups.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following inclusion criteria at the Screening and Baseline Visit (unless otherwise specified) to be eligible for inclusion in the SPIMD-301 trial:

1. Willing and able to provide a signed informed consent form (ICF) prior to participation in any trial-related procedures.
2. Agrees and is able to adhere to the trial requirements for the length of the trial, including administration of assigned treatment.
3. Is ≥18 years and ≤ 70 years of age at the time of screening.
4. Diagnosed with nPMD with a predominant clinical manifestation of myopathy, which must include progressive external ophthalmoplegia (PEO) and exercise intolerance and/or skeletal muscle weakness, with genetic confirmation of either:

   1. Nuclear DNA mutation of the mitochondrial replisome (replisome-related mutations), which include the following genes:

      * POLG 1/2
      * TWINKLE (C10ORF2)
      * TYMP
      * DGUOK
      * TK2
      * RRM2B
      * RNASEH1
      * SSBP
      * MGME1
      * DNA2
      * ANT1 (SLC25A4)
      * SUCLG1
      * SUCLA2
      * MPV17 or
   2. Other pathogenic mutations specific to nuclear DNA.
5. Women of childbearing potential must agree to use one of the following methods of birth control from the date they sign the ICF until 28 days after the last dose of IMP:

   1. Abstinence, when it is in line with the preferred and usual lifestyle of the subject. Subject agrees to use a highly effective method of contraception should they become sexually active.
   2. Relationships with male partners who have been surgically sterilized by vasectomy (the vasectomy procedure must have been conducted at least 60 days prior to the Screening Visit).
   3. Barrier method (e.g., condom or occlusive cap) with spermicidal foam/gel/film/cream AND either hormonal contraception (oral, implanted, or injectable) or an intrauterine device or system.

   Note: Non-childbearing potential is defined as surgical sterilization (e.g., bilateral oophorectomy, hysterectomy, or tubal ligation) or postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to the Screening Visit).
6. Male subjects with female partners of childbearing potential must be willing to use a highly effective method of contraception from the date they sign the ICF until 28 days after the last dose of IMP.

Exclusion Criteria:

1. Is unable to perform the 6MWT, 3TUG, or 5XSST functional tests. The use of a gait assist device is allowed; however, use should remain consistent for the entire duration of the trial.
2. Female subjects who are pregnant, planning to become pregnant, or breastfeeding/lactating.
3. Walks < 150 meters or > 450 meters during the 6MWT (Screening Visit only).
4. The estimated glomerular filtration rate (eGFR) is < 30 mL/min/1.73 m2, using the Modification of Diet in Renal Disease (MDRD) Study equation (Screening Visit only).
5. Has undergone an in-patient hospitalization within 30 days prior to screening or has a planned hospitalization or a surgical procedure during the trial, unless, in the opinion of the Investigator, it is concluded that it will not impact the outcome measurements of the trial.
6. Has clinically significant respiratory disease and/or cardiac disease that would interfere with trial assessments, in the opinion of the Investigator.
7. Has had any prior interventional cardiac procedure (e.g., cardiac catheterization, angioplasty/percutaneous coronary intervention, balloon valvuloplasty, etc.) within 3 months prior to screening.
8. Has history of or current severe neurologic impairment, severe epilepsy, severe ataxia, or severe neuropathy that may interfere with their ability to complete all trial requirements, in the opinion of the Investigator.
9. Active malignancy or any other cancer from which the subject has been disease-free for < 2 years. Localized squamous or non-invasive basal cell skin carcinomas are allowed, if appropriately treated prior to screening.
10. Has had a solid organ transplant.
11. Has been previously diagnosed with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
12. Has a history of a systemic eosinophilic illness and/or an eosinophil count >1,000 cells x106/L at the Screening Visit.
13. Is currently participating or has participated in an interventional clinical trial (i.e., investigational product or device, stem cell therapy, gene therapy) within 30 days prior to current trial; or is currently enrolled in a non-interventional clinical trial that, in the opinion of the Investigator, may be potentially confounding to the results of the current trial (e.g., exercise therapy trial).
14. Has received elamipretide (MTP-131) within the past one year of the Screening Visit.
15. Has a history of active substance abuse during the year prior, in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test (6MWT) | Baseline, Weeks 12, 24, 36, 48, 52 (End of Trial Visit)
  Change from Baseline in Distance Walked (in meters) on the Six-Minute Walk Test by Visit

SECONDARY OUTCOMES:
5 times sit-to-stand test (5XSST) | Baseline, Weeks 12, 24, 36, 48, 52 (End of Trial Visit)
  Change from Baseline in Total time (in seconds) to complete the 5XSST. Participant is directed to stand up straight as quickly as possible 5 times, without stopping in between, keeping arms folded across the chest. An average time is calculated.
Triple Timed up-and-go test (3TUG) | Baseline, Weeks 12, 24, 36, 48, 52 (End of Trial Visit)
  Change from Baseline in Total time (in seconds) to complete the 3TUG. Participant is directed to stand up from chair, walk at normal pace to the line on the floor 3 meters away, turn, walk back to the chair at normal pace, sit down again; activity is timed, in seconds. Activity is repeated 3 times consecutively without rest and an average time is calculated.
Patient Global Impression of Severity (PGI-S) Scale | Baseline, Weeks 12, 24, 36, 48
  Change from Baseline for PGI of Severity (PGI-S) Scale. Patient-reported current health status by week and at end of treatment. PGI-S Scale is a categorical scale and asks the participant to "rate the severity of your muscle weakness symptoms today" as one of the following categories: None, Mild, Moderate, Severe, or Very Severe. None means better health status, and best outcome, Very severe means worse health status and worse outcome.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (9):
  - University of California, San Diego, San Diego, California
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center College of Physician and Surgeon, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine Children's Hospital of Pittsburgh of UPMC Department of Genetics, Pittsburgh, Pennsylvania
  - UT Health,Center for the Treatment of Pediatric Neurodegenerative Disease, Houston, Texas
- Australia (2):
  - Royal North Shore Hospital Neurology, Sydney, New South Wales
  - Calvary Health Care Bethlehem, Parkdale, Victoria
- Germany (3):
  - Department of Neurology, University Clinics Munich, Munich, Bavaria
  - Universitaetsklinikum Carl Gustav Carus Dresden Neurologie, Dresden
  - Univ of Tubingen, Hertie Institute for Clinical Brain Research, Tübingen
- Hungary (2):
  - Semmelweis Egyetem Genomikai Medicina es Ritka Betegsegek, Budapest
  - University of Pécs, Department of Neurology Klinikai Kozpont - neurologiai Klinika, Pécs
- Italy (6):
  - University of Brescia, NeMO Clinical Center for Neuromuscular Diseases, Gussago, Brescia
  - Istituto di Neurologia, Fondazione Policlinico Universitario A. Gemelli, Università Cattolica del Sacro Cuore, Rome, Lazio
  - IRCCS Institute of Neorological Sciences of Bologna Bellaria Hospital, Bologna
  - Azienda Ospedaliero Universitaria Policlinico G. Martino, Messina
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Azienda Ospedaliero Universitario Pisana, Dipartimento Ambientale di Neuroscienze, Pisa
- Radboud University Medical Center, Nijmegen, Netherlands
- University of Auckland - Auckland City Hospital, Neurology Department, Auckland, New Zealand
- Helse Bergen HF, Bergen, Norway
- Spain (4):
  - Hospital de la Sta Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital la Fe de Valencia, Valencia
- United Kingdom (3):
  - University of Cambridge, Department of Clinical Neurosciences, Cambridge
  - Queen Square Centre for Neuromuscular Diseases The National Hospital for Neurology and Neurosurgery, London
  - Newcastle upon Tyne Hospitals Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No